CLINICAL TRIAL: NCT04871373
Title: The Effect of Motivational Interviewing on Oral Hygiene Behavior in Patients With Fixed Orthodontic Appliances: A Randomised Clinical Trial
Brief Title: Motivational Interview and Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Iberoamericana (Other)
Collaborators: Laboratorios Collado (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEI2017-06
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Motivational Interviewing; Oral Hygiene; Orthodontic Appliance Complication
Keywords: Motivational interviewing; Oral hygiene; Fixed orthodontic appliances; Treatment adherence
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Orthodontic patients were recruited to be divided into a control group (that received oral hygiene instructions) and an experimental group (that received oral hygiene instructions and motivational interviewing sessions).
Who Masked: Participant, Outcomes Assessor
Masking Description: Two dentists were in charge of the study logistic. They enrolled and allocated the participants according to the order of arrival and following the list of random numbers. A coding system was used as a concealment mechanism, which consisted of colored labels attached to the participants' file. This system was only known by the logistics managers and the interviewer (the periodontist who provided the OHI and the MI). Thus, the participant and the evaluator (the periodontist who recorded the data) were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A trained periodontist delivered oral hygiene instructions and motivational interviewing sessions. All the participants received a G.U.M. kit with special orthodontic hygiene tools.
  Interventions: Behavioral: Motivational interviewing; Behavioral: Oral Hygiene Instructions
- Control group (Active Comparator): A trained periodontist delivered only oral hygiene instructions. All the participants received a G.U.M. kit with special orthodontic hygiene tools.
  Interventions: Behavioral: Oral Hygiene Instructions

INTERVENTIONS:
Behavioral: Motivational interviewing — A periodontist was trained and evaluated by two expert psychologists in MI, who also supervised the interviewer to ensure that the intervention was properly applied. The periodontist conducted sessions of motivational interviewing monthly to the participants of the experimental group.
  Other Names: Motivational interview
  Arms: Experimental group
Behavioral: Oral Hygiene Instructions — A periodontist delivered OHI to all the participants of both studied groups. Also, every single patient received a G.U.M. kit with special orthodontic hygiene tools.
  Other Names: OHI

SUMMARY:
A parallel-group randomized clinical trial was conducted with 45 patients of the Orthodontic Clinic of Universidad Iberoamericana's (UNIBE) Postgraduate Unit. The study hypothesis was that motivational interview plus oral hygiene instructions would be more effective in maintaining long-term oral hygiene in comparison with conventional oral hygiene instructions alone.

A computer-generated list of numbers created with Statistical Package for the Social Sciences (SPSS) V21.0 was used to random allocate participants into the experimental or the control group. Monthly oral hygiene instructions and a G.U.M. kit were given to the sample. Additionally, the experimental group received motivational interviewing sessions by a trained periodontist. Simplified Oral Hygiene Index, Gingival Index, Periodontal Probing Depth and Bleeding on Probing were recorded at baseline, three and six months after the beginning of the study. Repeated-measures analysis of variance and chi-squared test were conducted.

DETAILED DESCRIPTION:
Sample calculation A power analysis was carried out to determine the number of subjects needed to achieve a Simplified Oral Hygiene Index (SOHI) significant interaction with the study groups when applying repeated measures ANOVA. The total number of completed subjects needed to achieve power of 0.90 with an alpha (α) of 0.05, an effect size (f) of at least .25 was determined to be 36; taking into consideration a possible 10% attrition rate, 45 subjects were recruited, consented and randomized to either the experimental or control group.

Due to the matter that repeated measures ANOVA treats each measurement as a separate variable, and it's preferable to use listwise deletion, if one measurement is missing, the whole case gets dropped. For this reason and therefore the incontrovertible fact that the trial suffers attrition, the sample for the three measurements was reduced to 32 subjects.

Randomization A simple randomization procedure was executed by the principal investigator to allocate the participants into one of the study groups. A computer-generated list of numbers was created using the software SPSS V21.0, with a 1:1.25 allocation ratio.

Two dentists enrolled and allocated the participants according to the order of arrival and following the list of random numbers. A coding system was used as a concealment mechanism, which consisted of colored labels attached to the participants' file. Thus, the participant and the evaluator (the periodontist who recorded the data) were masked.

Study intervention An interviewer was in charge of providing oral hygiene instructions for both groups. All the participants received a G.U.M. kit with special orthodontic hygiene tools. Then, the patients of the experimental group received a motivational interviewing session.

Afterward, the clinical parameters were measured by another periodontist. Monthly follow-up appointments were scheduled for the orthodontic check-ups to deliver a new G.U.M. kit, to reinforce the OHI and MI, and to register the periodontal parameters. The important data for this research was the one recorded at baseline, three and six months after the intervention.

Statistical analysis Mean Simplify oral hygiene index (SOHI), gingival index (GI), periodontal probing depth (PPD), and bleeding on probing (BoP) scores were compared between groups across three-time points using repeated-measures mixed-model analysis of variance. Tests for equality of variances and sphericity to check for homoscedasticity were performed due to the problem of sample attrition. Nevertheless, it was not found any violation to these assumptions in any of the variables included in the analysis. SPSS software was used for all calculations (IBM SPSS 25th version). Due to the nominal level of measurement of the variable BoP, it was performed a chi-squared test for each three time points to check if there were any differences between the two experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18-40 years old, systemically healthy, without active dental caries lesions or periodontal diseases, who were candidates for fixed orthodontic appliances.

Exclusion Criteria:

* Smokers and pregnant patients.
* Participants were discarded if they decided voluntarily to abandon the study of the orthodontic treatment or if they didn't attend to the periodical check-ups.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Simplified Oral Hygiene Index | Base line.
  six surfaces (from fou r posterior and two anterior teeth ) are examined for debris and calculus, whereas 12 surfaces are examined.
Simplified Oral Hygiene Index | 3rd month
  six surfaces (from fou r posterior and two anterior teeth ) are examined for debris and calculus, whereas 12 surfaces are examined.
Simplified Oral Hygiene Index | 6th month
  six surfaces (from fou r posterior and two anterior teeth ) are examined for debris and calculus, whereas 12 surfaces are examined.

SECONDARY OUTCOMES:
Gingival Index | Base line, 3 and 6 months after the intervention.
  Each of the four gingival areas of the tooth is given a score from 0 to 3; this is the gingival índex for the area.
Periodontal Probing Depth | Base line, 3 and 6 months after the intervention.
  One tooth per sextant was chosen and the average was calculated.
Bleeding on Probing | Base line, 3 and 6 months after the intervention.
  Dichotomic response after probing the gingival sulcus.

CONTACTS AND LOCATIONS:
Overall Officials: Henry A Adames, MsC, Principal Investigator — Universidad Iberoamericana
Locations (1):
- Universidad Iberoamericana UNIBE, Santo Domingo, Nacional, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yavan MA, Kocahan S, Ozdemir S, Sokucu O. The Effects of Using Plaque-Disclosing Tablets on the Removal of Plaque and Gingival Status of Orthodontic Patients. Turk J Orthod. 2019 Dec 1;32(4):207-214. doi: 10.5152/TurkJOrthod.2019.18084. eCollection 2019 Dec. PMID 32110465
- [Background] Alstad S, Zachrisson BU. Longitudinal study of periodontal condition associated with orthodontic treatment in adolescents. Am J Orthod. 1979 Sep;76(3):277-86. doi: 10.1016/0002-9416(79)90024-1. No abstract available. PMID 290273
- [Background] Petrauskiene S, Wanczewska N, Slabsinskiene E, Zemgulyte G. Self-Reported Changes in Oral Hygiene Habits among Adolescents Receiving Orthodontic Treatment. Dent J (Basel). 2019 Oct 1;7(4):96. doi: 10.3390/dj7040096. PMID 31581420
- [Background] Arici S, Alkan A, Arici N. Comparison of different toothbrushing protocols in poor-toothbrushing orthodontic patients. Eur J Orthod. 2007 Oct;29(5):488-92. doi: 10.1093/ejo/cjm038. PMID 17974538
- [Background] Moshkelgosha V, Mehrvarz S, Saki M, Golkari A. Computer-Based Oral Hygiene Instruction versus Verbal Method in Fixed Orthodontic Patients. J Dent Biomater. 2017 Mar;4(1):353-360. PMID 28959765
- [Background] Ousehal L, Lazrak L, Es-Said R, Hamdoune H, Elquars F, Khadija A. Evaluation of dental plaque control in patients wearing fixed orthodontic appliances: a clinical study. Int Orthod. 2011 Mar;9(1):140-55. doi: 10.1016/j.ortho.2010.12.013. Epub 2011 Feb 1. English, French. PMID 21277846
- [Background] Huang J, Yao Y, Jiang J, Li C. Effects of motivational methods on oral hygiene of orthodontic patients: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Nov;97(47):e13182. doi: 10.1097/MD.0000000000013182. PMID 30461616
- [Background] Skidmore KJ, Brook KJ, Thomson WM, Harding WJ. Factors influencing treatment time in orthodontic patients. Am J Orthod Dentofacial Orthop. 2006 Feb;129(2):230-8. doi: 10.1016/j.ajodo.2005.10.003. PMID 16473715
- [Background] Kay E, Locker D. A systematic review of the effectiveness of health promotion aimed at improving oral health. Community Dent Health. 1998 Sep;15(3):132-44. PMID 10645682
- [Background] Rollnick S, Miller WR, Butler C. Motivational Interviewing in Health Care. Helping Patients Change Behavior. New York, NY, USA: Guilford Press; 2008
- [Background] Miller WR, Rollnick S. Ten things that motivational interviewing is not. Behav Cogn Psychother. 2009 Mar;37(2):129-40. doi: 10.1017/S1352465809005128. PMID 19364414
- [Background] Gao X, Lo EC, McGrath C, Ho SM. Face-to-face individual counseling and online group motivational interviewing in improving oral health: study protocol for a randomized controlled trial. Trials. 2015 Sep 18;16:416. doi: 10.1186/s13063-015-0946-0. PMID 26385340
- [Background] Miller WR, Rollnick S. Motivational interviewing: Helping people change. 3rd ed. New York: Guilford Press; 2013
- [Background] Miller RW, Rollnick S. Motivational Interviewing: Preparing People for Change. New York: Guilford Press; 2002.
- [Background] Miller WR. A small study of training in motivational interviewing: does one workshop change clinician and client behavior? Behav Cogn Psychother 2001;29:457-71.
- [Background] Chen SM, Creedy D, Lin HS, Wollin J. Effects of motivational interviewing intervention on self-management, psychological and glycemic outcomes in type 2 diabetes: a randomized controlled trial. Int J Nurs Stud. 2012 Jun;49(6):637-44. doi: 10.1016/j.ijnurstu.2011.11.011. Epub 2011 Dec 30. PMID 22209215
- [Background] Koerber A, Crawford J, O'Connell K. The effects of teaching dental students brief motivational interviewing for smoking-cessation counseling: a pilot study. J Dent Educ. 2003 Apr;67(4):439-47. PMID 12749573
- [Background] Spirito A, Sindelar-Manning H, Colby SM, Barnett NP, Lewander W, Rohsenow DJ, Monti PM. Individual and family motivational interventions for alcohol-positive adolescents treated in an emergency department: results of a randomized clinical trial. Arch Pediatr Adolesc Med. 2011 Mar;165(3):269-74. doi: 10.1001/archpediatrics.2010.296. PMID 21383276
- [Background] Tripp SB, Perry JT, Romney S, Blood-Siegfried J. Providers as weight coaches: using practice guides and motivational interview to treat obesity in the pediatric office. J Pediatr Nurs. 2011 Oct;26(5):474-9. doi: 10.1016/j.pedn.2011.07.009. PMID 21930034
- [Background] Miller WR, Rose GS. Toward a theory of motivational interviewing. Am Psychol. 2009 Sep;64(6):527-37. doi: 10.1037/a0016830. PMID 19739882
- [Background] Tonetti MS, Eickholz P, Loos BG, Papapanou P, van der Velden U, Armitage G, Bouchard P, Deinzer R, Dietrich T, Hughes F, Kocher T, Lang NP, Lopez R, Needleman I, Newton T, Nibali L, Pretzl B, Ramseier C, Sanz-Sanchez I, Schlagenhauf U, Suvan JE. Principles in prevention of periodontal diseases: Consensus report of group 1 of the 11th European Workshop on Periodontology on effective prevention of periodontal and peri-implant diseases. J Clin Periodontol. 2015 Apr;42 Suppl 16:S5-11. doi: 10.1111/jcpe.12368. PMID 25639948
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Result] Rigau-Gay MM, Claver-Garrido E, Benet M, Lusilla-Palacios P, Ustrell-Torrent JM. Effectiveness of motivational interviewing to improve oral hygiene in orthodontic patients: A randomized controlled trial. J Health Psychol. 2020 Nov-Dec;25(13-14):2362-2373. doi: 10.1177/1359105318793719. Epub 2018 Sep 10. PMID 30198774
- [Result] Madariaga ACP, Bucci R, Rongo R, Simeon V, D'Anto V, Valletta R. Impact of Fixed Orthodontic Appliance and Clear Aligners on the Periodontal Health: A Prospective Clinical Study. Dent J (Basel). 2020 Jan 2;8(1):4. doi: 10.3390/dj8010004. PMID 31906577
- [Result] Gao X, Lo EC, Kot SC, Chan KC. Motivational interviewing in improving oral health: a systematic review of randomized controlled trials. J Periodontol. 2014 Mar;85(3):426-37. doi: 10.1902/jop.2013.130205. Epub 2013 Jun 27. PMID 23805818
- [Result] McGrath C. Behavioral Sciences in the Promotion of Oral Health. J Dent Res. 2019 Dec;98(13):1418-1424. doi: 10.1177/0022034519873842. PMID 31746683
- [Result] Renz A, Ide M, Newton T, Robinson PG, Smith D. Psychological interventions to improve adherence to oral hygiene instructions in adults with periodontal diseases. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD005097. doi: 10.1002/14651858.CD005097.pub2. PMID 17443571
- [Result] Brand VS, Bray KK, MacNeill S, Catley D, Williams K. Impact of single-session motivational interviewing on clinical outcomes following periodontal maintenance therapy. Int J Dent Hyg. 2013 May;11(2):134-41. doi: 10.1111/idh.12012. Epub 2012 Dec 24. PMID 23279918
- [Result] Kay EJ, Vascott D, Hocking A, Nield H. Motivational interviewing in general dental practice: A review of the evidence. Br Dent J. 2016 Dec 16;221(12):785-791. doi: 10.1038/sj.bdj.2016.952. PMID 27982007
- [Result] Cascaes AM, Bielemann RM, Clark VL, Barros AJ. Effectiveness of motivational interviewing at improving oral health: a systematic review. Rev Saude Publica. 2014 Feb;48(1):142-53. doi: 10.1590/s0034-8910.2014048004616. PMID 24789647
- [Result] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Result] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Result] Raju PK, Vasanti D, Kumar JR, Niranjani K, Kumar MS. Oral Hygiene Levels in Children of Tribal Population of Eastern Ghats: An Epidemiological Study. J Int Oral Health. 2015 Jul;7(7):108-10. PMID 26229382
- [Result] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Result] Chapple ILC, Mealey BL, Van Dyke TE, Bartold PM, Dommisch H, Eickholz P, Geisinger ML, Genco RJ, Glogauer M, Goldstein M, Griffin TJ, Holmstrup P, Johnson GK, Kapila Y, Lang NP, Meyle J, Murakami S, Plemons J, Romito GA, Shapira L, Tatakis DN, Teughels W, Trombelli L, Walter C, Wimmer G, Xenoudi P, Yoshie H. Periodontal health and gingival diseases and conditions on an intact and a reduced periodontium: Consensus report of workgroup 1 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S74-S84. doi: 10.1002/JPER.17-0719. PMID 29926944
- [Result] Discepoli N, Mirra R, Marruganti C, Beneforti C, Doldo T. Efficacy of Behaviour Change Techniques to improve oral hygiene control of individuals undergoing orthodontic therapy. A systematic review. Int J Dent Hyg. 2021 Feb;19(1):3-17. doi: 10.1111/idh.12468. Epub 2020 Oct 15. PMID 32974991
- [Result] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Result] Borrelli B, Tooley EM, Scott-Sheldon LA. Motivational Interviewing for Parent-child Health Interventions: A Systematic Review and Meta-Analysis. Pediatr Dent. 2015 May-Jun;37(3):254-65. PMID 26063554
- [Result] Stenman J, Wennstrom JL, Abrahamsson KH. A brief motivational interviewing as an adjunct to periodontal therapy-A potential tool to reduce relapse in oral hygiene behaviours. A three-year study. Int J Dent Hyg. 2018 May;16(2):298-304. doi: 10.1111/idh.12308. Epub 2017 Aug 24. PMID 28836375
- [Result] Faustino-Silva DD, Meyer E, Hugo FN, Hilgert JB. Effectiveness of Motivational Interviewing Training for Primary Care Dentists and Dental Health Technicians: Results from a Community Clinical Trial. J Dent Educ. 2019 May;83(5):585-594. doi: 10.21815/JDE.019.063. Epub 2019 Mar 11. PMID 30858274
- [Result] Moyers TB, Rowell LN, Manuel JK, Ernst D, Houck JM. The Motivational Interviewing Treatment Integrity Code (MITI 4): Rationale, Preliminary Reliability and Validity. J Subst Abuse Treat. 2016 Jun;65:36-42. doi: 10.1016/j.jsat.2016.01.001. Epub 2016 Jan 13. PMID 26874558
- [Result] Lundahl B, Burke BL. The effectiveness and applicability of motivational interviewing: a practice-friendly review of four meta-analyses. J Clin Psychol. 2009 Nov;65(11):1232-45. doi: 10.1002/jclp.20638. PMID 19739205
- [Result] Lundahl B, Droubay BA, Burke B, Butters RP, Nelford K, Hardy C, Keovongsa K, Bowles M. Motivational interviewing adherence tools: A scoping review investigating content validity. Patient Educ Couns. 2019 Dec;102(12):2145-2155. doi: 10.1016/j.pec.2019.07.003. Epub 2019 Jul 25. PMID 31514978

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04871373/Prot_SAP_000.pdf